CLINICAL TRIAL: NCT01343212
Title: Clinical Applications of Acoustic Radiation Force Impulse Technology in Stiffness Measurement of Liver Tumors and Visceral Parenchyma
Brief Title: Stiffness Measurement of Liver Tumors and Visceral Parenchyma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sheng-Hung Chen, China Medical University Hospital
Other Study IDs: DMR100-IRB-055
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; stiffness
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- newly diagnosed HCC: * Subjects with newly diagnosed untreated hepatocellular carcinoma (HCC) will be enrolled.
  * Subjects with the following conditions will be excluded:
  liver cancer other than HCC, treated HCC, post major abdominal surgery, contraindications to liver tumor biopsy, contraindications to local percutaneous treatment of liver tumors, low quality ARFI measurement
  Interventions: Other: stiffness measurement using ARFI

INTERVENTIONS:
Other: stiffness measurement using ARFI — Stiffness measurement will be performed for HCC using ARFI technique.
  Other Names: Acuson S2000

SUMMARY:
The investigators are measuring hepatocellular carcinoma(HCC)stiffness using Acoustic Radiation Force Impulse (ARFI) technique to enhance the diagnostic accuracy for HCC stratifications and treatment efficacy.

DETAILED DESCRIPTION:
Regression modelings as well as validity testings including cut-off identification will be acquired by performing both qualitative and quantitative measurements of HCC using reference diagnostic modalities e.g. pathology grading, dynamic CT scanning, etc.

ELIGIBILITY:
Inclusion Criteria:

with HCC

Exclusion Criteria:

* subjects with liver cancer other than HCC
* subjects with treated HCC
* post major abdominal surgery
* contraindications to liver tumor biopsy
* contraindications to local percutaneous treatment of liver tumors
* ARFI measurement low quality

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects with hepatocellular carcinoma(HCC)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Hung Chen, MD, Principal Investigator — Hepatogastroenterology, Department of Internal Medicine, China Medical University Hospital; Cheng-Yuan Peng, MD,PhD, Study Director — Hepatogastroenterology, Department of Internal Medicine, China Medical University Hospital
Locations (1):
- Hepatogastroenterology, Department of Internal Medicine, China Medical University Hospital, Taichung, Taiwan